CLINICAL TRIAL: NCT03154346
Title: Project Baseline Health Study
Status: Active, not recruiting | Type: Observational
Sponsor: Baseline Study LLC (Industry)
Collaborators: Verily Life Sciences LLC (Industry); Duke University (Other); Stanford University (Other); Google LLC. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-BL-001
Record Dates: First submitted 2017-04-19; First posted 2017-05-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: All
Keywords: Baseline; Project Baseline; Baseline Study; Project Baseline Study; Health Study; Baseline Health Study
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General Population: An unlimited number of participants will be accepted into a Baseline registry. From the Baseline registry, approximately 10,000 participants will be selected for the Baseline Study. Participant enrollment for the Baseline Study will be stratified by age, sex and risk factors and will aim to reflect the race and ethnicity distribution within the U.S.. The population includes a broad range of participants across the health spectrum, including exceptionally healthy participants, participants at risk of disease, and participants with current disease. The study population will be enriched for participants with an elevated risk of primary cardiovascular disease, lung cancer, and/or breast/ovarian cancers.

SUMMARY:
This study is the first initiative of Project Baseline, a broader effort designed to develop a well-defined reference, or "baseline," of good health as well as a rich data platform that may be used to better understand the transition from health to disease and identify additional risk factors for disease. Project Baseline endeavors to test and develop new tools and technologies to collect, organize, and activate health information.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* U.S. Resident
* Able to speak and read English
* Willing and able to comply with all aspects of the protocol

Exclusion Criteria:

* Individuals working on Project Baseline, including the Baseline Study
* Known severe allergy to nickel or metal jewelry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Project Baseline study population will be composed of adults across the health spectrum, including exceptionally healthy participants, participants at risk of disease, and participants with current disease.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-03-29 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Develop a set of scalable and standardized tools for acquiring, organizing, and analyzing clinical, molecular, imaging, sensor, self-reported, behavioral, environmental, and other health-related measurements | For the duration of the study
Evaluate the use of sensor technologies for the collection of continuous, accurate health information | For the duration of the study
Create a dataset encompassing a wide spectrum of phenotypic measures for future exploratory analysis | For the duration of the study
Measure the phenotypic diversity observed among a participant population, defining a range of expected values for multiple types of data | For the duration of the study
Identify biomarkers of disease-related transitions, including those related to cardiovascular disease and cancer | For the duration of the study

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Baseline Study, South San Francisco, California
  - Stanford Medicine, Stanford, California
  - California Health and Longevity Institute, Westlake Village, California
  - Duke University School of Medicine, Durham, North Carolina
  - Duke University School of Medicine, Kannapolis, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
It is envisioned that the Baseline Study data will be available to qualified researchers for exploratory analysis in the future. Qualified external researchers may apply through applications reviewed by the Proposal Review and Publications Committee and Scientific Executive Committee.

REFERENCES:
- [Derived] Carroll MK, Faheem S, Bouteiller J, Hernandez A, Mahaffey KW, Mega JL, Pagidipati N, Schaack T, Shah SH, Shashidhar S, Swope S, Williams D, Plowman RS, Simard EP, Short SA, Sullivan SS. Retention and characteristics associated with remote questionnaire completion in a general population cohort study: the project baseline health study. Front Digit Health. 2025 Jun 24;7:1520132. doi: 10.3389/fdgth.2025.1520132. eCollection 2025. PMID 40630050
- [Derived] Duran JM, Shrader P, Hong C, Haddad F, Santana EJ, Cauwenberghs N, Kouznetsova T, Salerno M, Bloomfield G, Koweek L, Hernandez A, Mahaffey KW, Shah SH, Douglas PS, Daubert MA; Project Baseline Health Study Group. Abnormal Exercise Electrocardiography With Normal Stress Echocardiography Is Associated With Subclinical Coronary Atherosclerosis. Circ Cardiovasc Imaging. 2025 Feb;18(2):e017380. doi: 10.1161/CIRCIMAGING.124.017380. Epub 2025 Jan 13. PMID 39801490
- [Derived] Feng KY, Short SA, Saeb S, Carroll MK, Olivier CB, Simard EP, Swope S, Williams D, Eckstrand J, Pagidipati N, Shah SH, Hernandez AF, Mahaffey KW. Resting Heart Rate and Associations With Clinical Measures From the Project Baseline Health Study: Observational Study. J Med Internet Res. 2024 Dec 20;26:e60493. doi: 10.2196/60493. PMID 39705694
- [Derived] Doroodgar Jorshery S, Chandra J, Walia AS, Stumiolo A, Corey K, Zekavat SM, Zinzuwadia AN, Patel K, Short S, Mega JL, Plowman RS, Pagidipati N, Sullivan SS, Mahaffey KW, Shah SH, Hernandez AF, Christiani D, Aerts HJWL, Weiss J, Lu MT, Raghu VK. Leveraging Deep Learning of Chest Radiograph Images to Identify Individuals at High Risk for Chronic Obstructive Pulmonary Disease. medRxiv [Preprint]. 2024 Nov 15:2024.11.14.24317055. doi: 10.1101/2024.11.14.24317055. PMID 39606360
- [Derived] Taylor KA, Carroll MK, Short SA, Celestin BE, Gilbertson A, Olivier CB, Haddad F, Cauwenberghs N. Factors associated with lower quarter performance-based balance and strength tests: a cross-sectional analysis from the project baseline health study. Front Sports Act Living. 2024 Jul 15;6:1393332. doi: 10.3389/fspor.2024.1393332. eCollection 2024. PMID 39081837
- [Derived] Kercheval JB, Narcisse DI, Nguyen M, Rao SV, Gutierrez JA, Leeper NJ, Maron DJ, Rodriguez F, Hernandez AF, Mahaffey KW, Shah SH, Swaminathan RV; Project Baseline Health Study Group. Characterization of peripheral artery disease and associations with traditional risk factors, mobility, and biomarkers in the project baseline health study. Am Heart J. 2024 Sep;275:183-190. doi: 10.1016/j.ahj.2024.06.010. Epub 2024 Jul 3. PMID 38969081
- [Derived] Uchehara B, Coulter Kwee L, Regan J, Chatterjee R, Eckstrand J, Swope S, Gold G, Schaack T, Douglas P, Mettu P, Haddad F, Shore S, Hernandez A, Mahaffey KW, Pagidipati N, Shah SH; Project Baseline Health Study Group. Accelerated Epigenetic Aging Is Associated With Multiple Cardiometabolic, Hematologic, and Renal Abnormalities: A Project Baseline Health Substudy. Circ Genom Precis Med. 2023 Jun;16(3):216-223. doi: 10.1161/CIRCGEN.122.003772. Epub 2023 Apr 11. PMID 37039013
- [Derived] Haddad F, Cauwenberghs N, Daubert MA, Kobayashi Y, Bloomfield GS, Fleischman D, Koweek L, Maron DJ, Rodriguez F, Liao YJ, Moneghetti K, Amsallem M, Mega J, Hernandez A, Califf R, Mahaffey KW, Shah SH, Kuznetsova T, Douglas PS; Project Baseline Health Study Investigators. Association of left ventricular diastolic function with coronary artery calcium score: A Project Baseline Health Study. J Cardiovasc Comput Tomogr. 2022 Nov-Dec;16(6):498-508. doi: 10.1016/j.jcct.2022.06.003. Epub 2022 Jul 5. PMID 35872137
- [Derived] Chatterjee R, Kwee LC, Pagidipati N, Koweek LH, Mettu PS, Haddad F, Maron DJ, Rodriguez F, Mega JL, Hernandez A, Mahaffey K, Palaniappan L, Shah SH; Project Baseline Health Study. Multi-dimensional characterization of prediabetes in the Project Baseline Health Study. Cardiovasc Diabetol. 2022 Jul 18;21(1):134. doi: 10.1186/s12933-022-01565-x. PMID 35850765
- [Derived] Califf RM, Wong C, Doraiswamy PM, Hong DS, Miller DP, Mega JL; Baseline Study Group. Biological and clinical correlates of the patient health questionnaire-9: exploratory cross-sectional analyses of the baseline health study. BMJ Open. 2022 Jan 4;12(1):e054741. doi: 10.1136/bmjopen-2021-054741. PMID 34983769